CLINICAL TRIAL: NCT03422380
Title: Energy Expenditure in Subjects Successful at Weight Loss Maintenance
Brief Title: Energy Expenditure and Weight Loss Maintenance
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 07-0584; 1K23DK078913 (NIH)
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Obesity; Weight Change, Body; Weight Loss; Physical Activity
Keywords: energy expenditure; adaptive thermogenesis; metabolic adaptation; weight loss maintenance
MeSH Terms: conditions — Obesity; Body Weight Changes; Weight Loss; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Weight Loss Maintainers (WLM): Individuals maintaining ≥13.6 kg (30 lb) weight loss for ≥1 year
- Normal Weight Controls (NC): Individuals with normal weight whose BMI was matched to the current BMI of the WLM. NC had to be weight stable and not maintaining a weight loss of ≥13.6kg
- Controls with Overweight/Obesity (OC): Individuals with overweight/obesity whose BMI was matched to the pre-weight loss maximum BMI of WLM. OC had to be weight stable and not maintaining a weight loss of ≥13.6kg

SUMMARY:
Obesity is reaching epidemic proportions and threatens both health and quality of life of people around the world. While many individuals succeed at short term weight loss, weight loss maintenance is the greatest barrier to successful treatment of obesity. High levels of physical activity are consistently associated with success in weight loss maintenance. The major goal of this proposal is to understand how and why high levels of physical activity are critical for long term maintenance of weight loss. This project takes advantage of the National Weight Control Registry (NWCR), which follows over 6000 individuals who have maintained a weight loss of ≥30 pounds for ≥1 year. Understanding how individuals successful at weight loss maintenance achieve energy balance will provide important insight into strategies to help more people sustain a weight loss.

DETAILED DESCRIPTION:
Participants were recruited in three groups: weight loss maintainers (WLM: maintaining ≥13.6 kg weight loss for ≥1 year), normal weight controls (NC: Body Mass Index (BMI) matched to current BMI of WLM), and controls with overweight/obesity (Overweight Controls (OC): BMI matched to pre-weight loss maximum BMI of WLM). The investigators hypothesize that total daily energy expenditure (TDEE) in WLM is similar to OC but is significantly higher then NC. High levels of volitional physical activity may compensate for the reduction in energy expenditure ("energy gap") that is the expected result of weight loss. This allows WLM to maintain a high level of "energy flux", which may facilitate optimal body weight regulation over time. The investigators will use doubly labeled water to compare TDEE in WLM and both NC and OC. The investigators will also compare individual components of TDEE including resting energy expenditure (REE), thermic effect of food (TEF), physical activity energy expenditure (PAEE), and physical activity level (PAL) between groups. The investigators also hypothesize that REE in WLM is similar to controls of both types under free living conditions, but will decrease following a period of physical inactivity and be significantly less than controls. Studies in rodents have consistently shown evidence of an increase in metabolic efficiency in the reduced obese state manifested by a lower than predicted REE. Studies in humans have shown mixed results, however few studies have controlled for habitual level of physical activity. Recent evidence suggests REE is greater in adults who perform regular exercise than their sedentary peers; this difference can be attributed in part to greater tonic sympathetic nervous system stimulation of REE that occurs in habitually exercising adults. The investigators believe there is an increase in metabolic efficiency in the reduced obese state manifested by a lower than predicted REE, and that high levels of physical activity function to "mask" or "correct" this metabolic efficiency. The investigators will compare REE under free living conditions and during an experimentally imposed period of reduced energy flux (restricted physical activity matched by an equivalent reduction in energy intake) in WLM and controls.

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* Age 18-65
* Weight stable (<10 lb fluctuation in body weight over previous 6 months) or
* NWCR subjects successful at weight loss maintenance (maintaining a loss of ≥ 30 pounds for at least 2 years)
* Non-Reduced Weight Matched Controls: Individuals matched to NWCR subjects' current body weight. These individuals will be normal weight (BMI 18-25, BMI up to 27 allowed in men with waist circumference < 40 cm), and have no history of overweight or obesity (BMI >25) and will not be maintaining a weight loss ≥ 30 pounds.
* Non-Reduced Obese Controls: Individuals matched to NWCR subjects' maximum pre-weight loss body weight. These individuals will be overweight or obese (BMI ≥ 26-45).

Exclusion Criteria:

* Diabetes
* Uncontrolled HTN (>160/100)
* History of cardiac disease: CHF or angina, atrial fibrillation or ventricular tachycardia, or significant abnormality on resting EKG
* Symptoms suggestive of cardiovascular disease: chest pain, shortness of breath at rest or with mild exertion, dizziness, syncope.
* History of neurological disease: stroke, TIA or seizure disorder
* Current treatment for cancer (except skin)
* Severe pulmonary, liver or kidney disease
* Untreated thyroid disorder
* Severe arthritis or other musculoskeletal disorder
* Alcohol or drug abuse
* Active psychiatric illness
* Positive response to PAR-Q indicating requirement for monitored physical activity
* Other serious medical condition as determined by the investigator which would limit physical activity or require monitored activity.
* Pregnant and lactating women, and women actively trying to become pregnant (post-menopausal women on a stable dose of HRT and pre-menopausal women on a stable OCP regimen will be allowed to participate)
* Smoking within the past 6 months
* Subjects using prescription or over the counter medication which may affect RMR including beta blockers, stimulants such as Ritalin and appetite suppressants.
* Subjects who have undergone bariatric surgery or who are currently maintaining their weight loss with prescription weight loss drugs or supplements.
* Severe claustrophobia
* Moderate or high levels of physical activity at the workplace and unable to reduce workplace activity, work from home or take time off from work to participate in Study 2.
* We will exclude controls if they are weight reduced (maintaining a weight loss of ≥ 30 pounds).

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The proposed study design is aimed at collecting additional data on previously enrolled adult study subjects in the NWCR, which does not include children. The NWCR contains approximately 70% women and 30% men. We anticipate studying equal numbers of men and women in this study. Minorities comprise approximately 7% of total subjects in the NWCR. In the proposed studies, there will be no exclusions for racial or ethnic background.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Total Daily Energy Expenditure (TDEE) | At 8 days
  After a 12-hour overnight fast, participants provided a baseline urine sample on day 1. Participants were then administered an oral dose of doubly labeled water (DLW) containing 1.8g 10% 18O/kg total body water (TBW) and 0.12 g/kg TBW of 99.9% deuterium. TBW was estimated as 73% of FFM from DXA. The dosing cup was rinsed twice with 30 mL of water and the rinsing dose consumed. Exact time of dosing was recorded. Additional urine samples were collected after a 4hr and 5hr post-dose equilibrium period and then again at the same times on day 8. TDEE over days 1-8 was determined using a single DLW dose and the two-point method according to Schoeller and colleagues.

SECONDARY OUTCOMES:
Physical Activity Energy Expenditure (PAEE) | At 8 days
  PAEE was calculated as TDEE - TEF - REE. In addition, because the energy cost of PA is proportional to body weight for a given intensity and duration, PAEE was also calculated as relative to body weight (kg).
Resting Energy Expenditure (REE) | Day 1 and Day 8 over a 1 week period
  REE was measured using standard indirect calorimetry (Truemax 2400, ParvoMedics, Salt Lake City, UT) with the ventilated hood technique. Study participants arrived at 7am after a 12-hour overnight fast. Participants rested supine, awake, and lightly clothed in a thermoneutral (68-74 ˚F), dimly lit, quite room for 30 minutes. Respiratory gas exchange was measured for 15 minutes, using the last 10 minutes to average REE. Tests were examined for validity to confirm a) average RQ was 0.7-0.9, and b) average Metabolic Equivalents (METs) <1.10. If the averaged data fell outside of these ranges, the test was considered invalid and excluded from the analysis. REE was collected on days 1 and 8 of the free-living monitoring period, and averaged to produce a single value for REE (intraclass correlation coefficient = 0.96).
Thermic Effect of Food (TEF) | At 8 days
  The thermic effect of food (TEF) was calculated as 10% of TDEE.
Physical Activity Level (PAL) | At 8 days
  PAL was calculated as TDEE/REE.

OTHER OUTCOMES:
Physical Activity Patterns | At 8 days
  PA patterns were assessed using the activPALTM activity monitor (PAL Technologies, Glasgow, Scotland). The activPALTM is a small (23x43x5 mm) and lightweight (10 grams) device that uses accelerometer-derived information about thigh position to estimate time spent sitting/lying, standing, and stepping. The device is attached to the anterior thigh and is waterproofed by wrapping it in a nitrile sleeve, allowing for 24-hour measurement. Participants were asked to wear the device continuously for seven days.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Catenacci, MD, Principal Investigator — University of CO
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

REFERENCES:
- [Derived] Dahle JH, Ostendorf DM, Zaman A, Pan Z, Melanson EL, Catenacci VA. Underreporting of energy intake in weight loss maintainers. Am J Clin Nutr. 2021 Jul 1;114(1):257-266. doi: 10.1093/ajcn/nqab012. PMID 33742193
- [Derived] Ostendorf DM, Caldwell AE, Creasy SA, Pan Z, Lyden K, Bergouignan A, MacLean PS, Wyatt HR, Hill JO, Melanson EL, Catenacci VA. Physical Activity Energy Expenditure and Total Daily Energy Expenditure in Successful Weight Loss Maintainers. Obesity (Silver Spring). 2019 Mar;27(3):496-504. doi: 10.1002/oby.22373. PMID 30801984
- [Derived] Ostendorf DM, Melanson EL, Caldwell AE, Creasy SA, Pan Z, MacLean PS, Wyatt HR, Hill JO, Catenacci VA. No consistent evidence of a disproportionately low resting energy expenditure in long-term successful weight-loss maintainers. Am J Clin Nutr. 2018 Oct 1;108(4):658-666. doi: 10.1093/ajcn/nqy179. PMID 30321282